CLINICAL TRIAL: NCT00422344
Title: A Phase I Study of RAD001 and Sunitinib in Metastatic Renal Cell Carcinoma Patients
Brief Title: A Study of RAD001 and Sunitinib in Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Glenn Kroog, MD, Memorial Sloan Kettering Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-105
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
Keywords: RAD001; Sunitinib; renal; kidney
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus; Sunitinib

ARMS (1):
- RAD001 AND SUNITINIB (Experimental): RAD001 AND SUNITINIB IN METASTATIC RENAL CELL CARCINOMA PATIENTS
  Interventions: Drug: RAD001, Sunitinib

INTERVENTIONS:
Drug: RAD001, Sunitinib — Patients will start treatment with Sunitinib and RAD001 on Cycle 1, Day 1. Sunitinib will be given orally daily for 4 weeks followed by a 2 week rest period. RAD001 will be given orally daily or weekly in subsequent cohorts with the first treatment on day 1. DLT determination will be based on toxicities observed in Cycles 1 - a cycle being defined by Sunitinib dosing. Once the MTD for the combination has been identified, a total of 10 patients will be enrolled into the study at the highest dose level that allows for administration of multiple cycles and provides potentially therapeutic drug levels of both drugs

SUMMARY:
The purpose of this study is to test the safety of RAD-001 and Sunitinib given in combination for renal cell cancer. We also want to find out what effects (good and bad) the combination of RAD-001 and Sunitinib have on you and your tumor.

RAD001 is a pill that works by shutting down some of the pathways in the cell that make tumors grow. Sunitinib is a pill that works by shutting off the signal in the cancer cells that tell the cells to grow blood vessels. Without this signal, the blood vessels to the tumors shrink down.

DETAILED DESCRIPTION:
To assess the maximum tolerated doses and overall safety and tolerability of Sunitinib administered in combination with RAD001 for the treatment of patients with metastatic renal cell carcinoma.

To assess antitumor activity of the combination of Sunitinib and RAD001.

This study is designed to confirm that the 2 agents can be administered safely in combination. Patients will begin treatment with Sunitinib and RAD001 on Day 1. RAD001 will be administered orally on a weekly schedule. Sunitinib will be given orally on a 4 weeks on, 2 weeks off schedule. DLT determination will be based on toxicities observed in Cycle 1 - a cycle is defined by Sunitinib dosing ( 6 weeks). Once the MTD for the combination has been identified, a total of 10 patients will be enrolled at the highest dose level that allows for administration of multiple cycles and provides potentially therapeutic drug levels of both drugs to further assess safety and tolerability and to obtain a preliminary assessment of efficacy. Patients will be treated with RAD001 and Sunitinib until there is disease progression, significant toxicity or withdrawal of patient consent. Patients judged to derive benefit from treatment would be offered participation in a continuation protocol at the conclusion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Any histologically confirmed renal cell carcinoma with metastases. Patients with unresected primary tumors may be enrolled as long as evidence of metastatic disease is also present.
* No prior sunitinib or m-TOR inhibitor. The washout period must be at least 4 weeks for any prior therapy.
* Male or female, 18 years of age or older.
* ECOG performance status 0 or 1.
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, or surgical procedure to NCI CTCAE grade less than or equal to 1.
* Adequate organ function as defined by the following criteria:
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) less than or equal to 2.5 x upper limit of normal (ULN) or less than 5 x ULN in the presence of liver metastases.
* Total serum bilirubin less than or equal to 1.5 mg/dL
* Total leukocyte count greater to or equal to 3000 cells/ul
* Absolute neutrophil count (ANC) greater than or equal to 1500/µL
* Platelets greater than or equal to 100,000/µL
* Hemoglobin greater than or equal to 9.0 g/dL
* Serum calcium less than or equal to 12.0 mg/dL
* Serum creatinine less than or equal to 2.0 x ULN
* PT less than or equal to 1.5 ULN
* Negative serum or urine pregnancy test in women of child-bearing age
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Major surgery, open biopsy, traumatic injury, radiation or systemic therapy within 4 weeks of starting the study treatment. Anticipation of major surgical procedure during the study. Prior palliative radiotherapy to metastatic lesion(s)is permitted, provided there is at least one measurable lesion that has not been irradiated.
* More than 3 prior systemic therapies for metastatic RCC.
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0.
* No other approved or investigational anticancer treatment will be permitted during the study period, including chemotherapy, biological response modifiers, hormone therapy, or immunotherapy, with the exception of palliative radiation therapy. No other investigational drug may be used during treatment on this protocol, and concurrent participation in another clinical trial is not allowed.
* NCI CTCAE grade 3 hemorrhage within the past 1 month.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
* Chronic treatment with systemic steroids or other immunosuppressive agent
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Sunitinib or RAD001 (e.g. malabsorptive disorder, ulcerative disease, uncontrolled nausea, vomiting, diarrhea, or small bowel resection)
* Patients with an active bleeding diathesis or on oral anti-vitamin K medication (except low dose warfarin)
* Current spinal cord compression, or carcinomatous meningitis.
* Any of the following within the 12 months prior to study drug administration:

  * severe/unstable angina,
  * MI,
  * CABG,
  * symptomatic congestive heart failure,
  * cerebrovascular accident or transient ischemic attack or peripheral vascular disease.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade greater or equal to 2, atrial fibrillation of any grade, or prolongation of the QTc interval to >450 msec for males and >470 msec for females.
* Blood pressure > 150/100mmHg
* Evidence of bleeding diathesis or coagulopathy
* Serious, non-healing wound, ulcer or bone fracture
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Current treatment on another therapeutic clinical trial.
* Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy.
* Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Receipt of any investigational agent within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated doses and overall safety and tolerability of Sunitinib administered in combination with RAD001 for the treatment of patients with metastatic renal cell carcinoma. | toxicities observed in Cycle 1 - a cycle is defined by Sunitinib dosing ( 6 weeks)

SECONDARY OUTCOMES:
To assess antitumor activity of the combination of Sunitinib and RAD001. | conclusion of this study

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Kroog, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org